CLINICAL TRIAL: NCT00413413
Title: A Multi-national, Multicenter, Double-blind, Double-dummy, Randomized, Active-controled, Parallel Study, Comparing Efficacy and Safety of Valsartan/Amlodipine 80/5 mg to Valsartan 80 mg and Valsartan 160 mg Alone Once Daily in Patients With Mild to Moderate Essential Hypertension Not Adequately Controlled With Valsartan 80 mg Monotherapy.
Brief Title: Efficacy/Safety of Valsartan Plus Amlodipine and Valsartan Alone in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2316
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2009-09-14 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: Hypertension, valsartan, amlodipine, high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Valsartan/amlodipine 80/5 mg (Experimental)
  Interventions: Drug: Valsartan/amlodipine 80/5 mg
- Valsartan 80 mg (Active Comparator)
  Interventions: Drug: Valsartan 80 mg
- Valsartan 160 mg (Active Comparator)
  Interventions: Drug: Valsartan 160 mg

INTERVENTIONS:
Drug: Valsartan/amlodipine 80/5 mg — 1 valsartan/amlodipine 80/5 mg tablet, 1 placebo capsule to match valsartan once daily
  Arms: Valsartan/amlodipine 80/5 mg
Drug: Valsartan 80 mg — 1 valsartan 80 mg capsule, 1 placebo tablet to match valsartan/amlodipine 80/5 mg once daily
  Arms: Valsartan 80 mg
Drug: Valsartan 160 mg — 1 valsartan 160 mg capsule, 1 placebo tablet to match valsartan/amlodipine 80/5 mg once daily
  Arms: Valsartan 160 mg

SUMMARY:
This study evaluated the safety and efficacy of the fixed combination of valsartan/amlodipine in adult patients with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients >= 18 years and < 86 years
* Patients with essential diastolic hypertension
* At visit 1, the patient must have mean sitting diastolic blood pressure >= 95 mmHg and < 10 mmHg; patients treated with antihypertensive medication must have a mean sitting diastolic blood pressure < 100 mmHg
* At visit 2, patients must have a mean sitting diastolic blood pressure of >= 95 mmHg and < 100 mmHg
* At visit 3, patients must have a mean sitting diastolic blood pressure of >= 90 mmHg and < 110 mmHg

Exclusion Criteria:

* Severe hypertension >= 180/110 mmHg
* Known or suspected contraindications, including a history of allergy or hypersensitivity to valsartan or amlodipine or to other drugs with similar chemical structures
* Inability to discontinue all prior antihypertensive medications safely for a maximum period of up to 28 days prior to Visit 2
* History of hypertensive encephalopathy, cerebrovascular accident or transient ischemic attack, myocardial infarction or other types of revascularization
* Malignant hypertension
* All patients with Type I diabetes and those patients with Type 2 diabetes who are not well controlled based on the investigator's clinical judgment
* Pregnant or nursing women
* History of heart failure
* Angina pectoris
* Second or third degree heart block
* Life threatening or symptomatic arrhythmias
* Clinically significant valvular heart disease
* Evidence of a secondary form of hypertension
* Known or moderate malignant retinopathy
* Evidence of hepatic disease
* Evidence of renal impairment

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1134 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- China (19):
  - Beijing ChaoYang Hospital, Affiliate of Capital University of Medical Sciences, Beijing
  - Beijing General Hospital of Beijing Military Region, Beijing
  - Beijing Hospital, Beijing
  - The First People's Hospital of Hangzhou, Hangzhou
  - The Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou
  - The First Affiliated Hospital of Medical College of Zhejiang University, Hangzhou
  - Southeast University Affiliated Zhong Da Hospital, Nanjing
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Second Military Medical University Affiliated Changzheng Hospital, Shanghai
  - Department of cardiology, Ruijin hospital;, Shanghai
  - Department of cardiology, Ruijin hospital, Shanghai
  - Fudan University affiliated zhongshan hospital, Shanghai
  - Second Military Medical University Affiliated Changhai Hospital, Shanghai
  - The First Affiliated Hospital of China Medical University, Shenyang
  - The people's Hospital of Liaoning Province, Shenyang
  - Second Hospital of Hebei University of Medical Sciences, Shijiazhuang
  - The People's Hospital of Hebei Provincial, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - The First Affiliated Hospital of Soochow University, Suzhou

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1134 patients were enrolled into the single-blind period of the study, and 216 (19%) were discontinued. In total, 918 patients were randomized to the three treatment groups.
Period: Single-Blind
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg
Started | 0 (In single-blind period participants were only enrolled to Valsartan 80 mg arm.) | 1134 | 0 (In single-blind period participants were only enrolled to Valsartan 80 mg arm.)
Completed | 0 | 918 | 0
Not Completed | 0 | 216 | 0
Not completed — Adverse Event | 0 | 9 | 0
Not completed — Lack of Efficacy | 0 | 5 | 0
Not completed — Subject no longer requires study drug | 0 | 151 | 0
Not completed — Protocol Violation | 0 | 16 | 0
Not completed — Withdrawal by Subject | 0 | 27 | 0
Not completed — Lost to Follow-up | 0 | 8 | 0
Period: Double-Blind
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg
Started | 308 | 307 | 303
Completed | 293 | 293 | 285
Not Completed | 15 | 14 | 18
Not completed — Adverse Event | 6 | 0 | 5
Not completed — Unsatisfactory therapeutic effect | 1 | 2 | 1
Not completed — Protocol deviation | 1 | 2 | 1
Not completed — Subject withdrew consent | 4 | 6 | 9
Not completed — Lost to Follow-up | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg | Total
Number analyzed (Participants) | 308 | 306 | 302 | 916
Age Continuous [Mean (Standard Deviation); unit: years] — All baseline measures were based on Full-set analysis population. Two patients were excluded from the full-set analysis population for having no post-baseline efficacy assessment. All randomized patients were included in the safety population.
  years | 51.6 (10.8) | 51.7 (8.9) | 51.2 (9.6) | 51.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 115 | 104 | 346
  Male | 181 | 191 | 198 | 570

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study (Week 8)
Description: Blood pressure (BP) was measured with a calibrated aneroid or mercury sphygmomanometer. The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position for five minutes, systolic/diastolic BP was measured 3 times at 1-2-minute intervals. The mean of the 3 measurements was calculated.
Time Frame: Baseline to end of study (Week 8)
Population: Full-set analysis population: All randomized patients who had a baseline and at least one post-baseline efficacy measurement. For patients who did not complete the Week 8 assessment, a last observation carried forward (LOCF) approach was used.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 308 | 306 | 302
mmHg | -10.8 (0.42) | -6.3 (0.42) | -7.2 (0.42)

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to End of Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: Full-set analysis population population: All randomized patients who had a baseline and at least one post-baseline efficacy measurement. For patients who did not complete the Week 8 assessment, a last observation carried forward (LOCF) approach was used.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 308 | 306 | 302
mmHg | -12.5 (0.61) | -6.0 (0.62) | -7.7 (0.62)

3. Secondary Outcome: Percentage of Patients Achieving a Diastolic Blood Pressure Response at the End of the Study (Week 8)
Description: A diastolic blood pressure response was defined as a msDBP < 90 mmHg or a ≥ 10 mmHg decrease compared to baseline at the end of the study (Week 8). Blood pressure (BP) was measured with a calibrated aneroid or mercury sphygmomanometer. The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position for five minutes, systolic/diastolic BP was measured 3 times at 1-2-minute intervals. The mean of the 3 measurements was calculated.
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 308 | 306 | 302
Percentage of patients | 77.9 | 57.8 | 66.6

4. Secondary Outcome: Percentage of Patients Achieving Diastolic Blood Pressure Control at the End of the Study (Week 8)
Description: Diastolic blood pressure control was defined as a msDBP < 90 mmHg at the end of the study (Week 8). Blood pressure (BP) was measured with a calibrated aneroid or mercury sphygmomanometer. The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position for five minutes, systolic/diastolic BP was measured 3 times at 1-2-minute intervals. The mean of the 3 measurements was calculated.
Time Frame: End of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 308 | 306 | 302
Percentage of patients | 74.4 | 53.6 | 64.2

5. Secondary Outcome: Percentage of Patients Achieving Overall Blood Pressure Control at the End of the Study (Week 8)
Description: Overall blood pressure control rate was defined as a msSBP/msDBP < 140/90 mmHg at the end of the study (Week 8). Blood pressure (BP) was measured with a calibrated aneroid or mercury sphygmomanometer. The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position for five minutes, systolic/diastolic BP was measured 3 times at 1-2-minute intervals. The mean of the 3 measurements was calculated.
Time Frame: End of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 308 | 306 | 302
Percentage of patients | 70.5 | 44.1 | 58.6

ADVERSE EVENTS:
Arm/Group | Valsartan/Amlodipine 80/5 mg | Valsartan 80 mg | Valsartan 160 mg
Serious Adverse Events (participants affected / at risk) | 4/308 | 0/307 | 4/303
Other Adverse Events (participants affected / at risk) | 0/308 | 0/307 | 0/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/Amlodipine 80/5 mg (N=308) | Valsartan 80 mg (N=307) | Valsartan 160 mg (N=303)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.